CLINICAL TRIAL: NCT02627079
Title: ICanSTEP: Increasing Physical Activity in Cancer Survivors Through a Text-messaging Exercise Motivation Program
Brief Title: ICanSTEP : Increasing Physical Activity With Text Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00068978
Record Dates: First submitted 2015-12-08; First posted 2015-12-10 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: A Diagnosis of Any Hematologic or Solid Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): Cohort 1 will include 15 sedentary participants who have completed all cancer therapy except adjuvant hormonal therapy.
  All participants will be provided a Fitbit. Participants will then be provided daily SMS text messaging tailored to their activity level for 12 weeks..
  Interventions: Other: Daily SMS text messaging
- Cohort 2 (Active Comparator): Cohort 2 will include 15 sedentary participants in active treatment. All participants will be provided a Fitbit. Participants will then be provided daily SMS text messaging tailored to their activity levels for 12 weeks.
  Interventions: Other: Daily SMS text messaging

INTERVENTIONS:
Other: Daily SMS text messaging

SUMMARY:
The proposed pilot study will develop and test feasibility and preliminary efficacy of an exercise motivation intervention using a 12-week smartphone-text messaging program tailored to physical activity data retrieved from a Fitbit. Target population is 15 cancer survivors and 15 patients actively undergoing cancer treatment.

DETAILED DESCRIPTION:
Cancer survivors have substantial residual cardiometabolic risk due to the fact that they are living longer and are exposed to the same lifestyle and environmental factors that have led to the drastic increase in obesity and diabetes in Western societies over the last four decades. In addition, survivors' cardiovascular health is significantly impaired due to cancer treatment. Research has shown that physical activity improves quality of life in cancer survivors, ameliorates treatment-related side effects reduces the risk of cancer recurrence, and extends overall survival. Despite these advantages, most cancer patients are sedentary. The early survivor period is a teachable moment to improve healthy behaviors. Social Cognitive Theory argues that to change exercise behavior, we must increase behavior change self-efficacy of participants (i.e., confidence), increase their outcome expectations that changing their behavior will lead to better health, enhance motivation to exercise, enhance their ability to regulate their behavior (self-regulation), teach them tangible behavior change skills, and help them overcome barriers to behavior change. In this study validated patient-reported outcomes will be performed at baseline and at 12 weeks - FACIT-F to document general cancer symptoms with additional questions on fatigue, the Beck Depression Inventory (BDI-II), and the modified Godin-Leisure Questionnaire as a measure of activity level. The investigators will also perform baseline and 3 month weight / BMI and 6-minute walk testing as a second well-validated objective measure of fitness. At enrollment and at 3 months, patients will be queried as to barriers to behavior change. At 3 months, patients will be asked by 5-point Likert scale how helpful the program was in increasing their physical activity. Six months after enrollment (+/- 4 weeks), level of physical activity and use of Fitbit will be determined.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants must be / have

1. age 18 or older,
2. a diagnosis of any hematologic or solid malignancy
3. a life expectancy of at least 12 months
4. ECOG < /=2
5. in active cancer treatment or have completed active cancer treatment within one year of obtaining consent (with the exception of adjuvant hormonal therapy),
6. not scheduled for any major surgery during the anticipated study period,
7. able to read and understand English
8. sedentary defined as participating in 2 or less days of dedicated physical activity per week,
9. consistent daily access to a smartphone
10. a text messaging plan that includes a minimum of 150 text messages a month at no additional cost
11. capable of providing informed consent.

Exclusion Criteria:

1. Significant cardiac disease (i.e., left ventricular ejection fraction of <50%, unstable angina, placement of cardiac stents and myocardial infarction within previous 6 months)
2. Contraindications to a 6-minute walk test as recommended by the American Thoracic Society: (a) acute myocardial infarction (3-5 days), (b) unstable angina, (c) uncontrolled arrhythmias causing symptoms or hemodynamic compromise, (d) syncope, (e) acute endocarditis, (f) acute myocarditis or pericarditis, (g) uncontrolled heart failure, (h) acute pulmonary embolus or pulmonary infarction, (i) thrombosis of lower extremities, (j) suspected dissecting aneurysm, (k) uncontrolled asthma, (l) pulmonary edema, (m) room air desaturation at rest ≤85%, (n) respiratory failure, (o) acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise, (p) mental impairment leading to inability to cooperate, and (q) extensive bone metastases
3. ECOG >2
4. Participates in 3 or more days of dedicated physical activity per week
5. Known allergic reaction to nickel
6. No access to a smart phone or text messaging plan less than 150 messages per month
7. Physical or psychological contraindication to participation at the discretion of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Feasibility, as measured by the percentage of eligible patients who can be enrolled | 6 months
Feasibility, as measured by accrual rate | 6 months
Change in daily step count, as measured by Fitbit | Baseline, 12 weeks
Change in minutes of weekly exercise, as measured by Fitbit | Baseline, 12 weeks
Change in fatigue, as measured by questionnaire | Baseline, 12 weeks
Change in depression, as measured by questionnaire | Baseline, 12 weeks
Change in general activity, as measured by questionnaire | Baseline, 6 months
Change in quality of life, as measured by questionnaire | Baseline, 12 weeks
Change in body mass index (BMI) | Baseline, 12 weeks

SECONDARY OUTCOMES:
Mean difference in daily step count, as measured by Fitbit | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.
Mean difference in minutes of weekly exercise, as measured by Fitbit | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.
Mean difference in fatigue, as measured by questionnaire | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.
Mean difference in depression, as measured by questionnaire | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.
Mean difference in general activity, as measured by questionnaire | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.
Mean difference in quality of life, as measured by questionnaire | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.
Mean difference in body mass index (BMI) | Baseline, 12 weeks
  This will be addressed by calculating the mean difference (with 80% confidence interval) between the two treatment cohorts in change across time.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Koontz, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koontz BF, Levine E, McSherry F, Niedzwiecki D, Sutton L, Dale T, Streicher M, Rushing C, Owen L, Kraus WE, Bennett G, Pollak KI. Increasing physical activity in Cancer Survivors through a Text-messaging Exercise motivation Program (ICanSTEP). Support Care Cancer. 2021 Dec;29(12):7339-7349. doi: 10.1007/s00520-021-06281-y. Epub 2021 May 28. PMID 34050402